CLINICAL TRIAL: NCT03428087
Title: Prostate Impendance Test Project (PROS.IT) in Prostate Cancer Diagnosis: a Cross-sectional Observational Study
Brief Title: Prostate Impendance Test Project
Acronym: PROSIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Riccardo Bartoletti, Prostate Impedance Test (PROS.iT) Project in prostate cancer diagnosis: a cross-sectional observational study, University of Pisa
Other Study IDs: 151/2016
Record Dates: First submitted 2018-02-03; First posted 2018-02-09 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Prostatic Neoplasms; PSA; Prostatic Biopsy; Impedance Test
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients undergoing prostatic biopsy: Patients who are candidates for prostate biopsy as suffering from urinary symptoms accompanied by clinical suspicions such as high total PSA value and / or presence of prostate nodule and / or evidence of obvious lesion to available imaging methods.

SUMMARY:
Impedance-based analysis could provide an adequate response to the need to identify a safe and reliable tool alternative to bioptic diagnosis. Patients who are candidates for prostate biopsy as suffering from urinary symptoms accompanied by clinical suspicions such as high total PSA value and / or presence of prostate nodule and / or evidence of obvious lesion to available imaging methods will be subjected to impedance measurement. Aim of this study is to be able to structure a bivariate analysis of the distribution of impedances detected in patients with neoplasia in order to detect test median reference values.

ELIGIBILITY:
Inclusion Criteria:

1. age> 45 years
2. up of total PSA values beyond the normal range (> 4 ng / ml)
3. presence or absence of suspicious prostate nodule

Exclusion Criteria:

1. previous history of cancer
2. BMI>30
3. patients with previous diagnosis of PIN HG at prostate core biopsy or in active surveillance

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In order to build a two-pronged analysis of areas of confidence and tolerance, it is necessary to examine a fair number of potentially ill subjects and compare them with healthy subjects (controls). Past experiences indicate that about 100 measurements in each grop can create a sufficiently dense and significant cluster to be able to trace besides the "boundries" of 50%, 75%, and 95% even a 95% confidence center of small size suitable to establish an adequate significance.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Impedance-based analysis based on phase-sensitive sensors | during rectal examination

CONTACTS AND LOCATIONS:
Locations (1):
- AOUP Ospedale cisanello, Pisa, Tuscany, Italy